CLINICAL TRIAL: NCT06807086
Title: Efficacy of Synchronous, Virtual Cognitive Behavioral Therapy for Insomnia Across Phases of Cancer Survivorship
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Daniel L Hall, PhD, Assistant Professor of Psychology, Associate Director of Utilization & Evaluation Research, Health Promotion & Resiliency Intervention Research Center, Psychologist, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSG-24-1247084-01-CTPS
Record Dates: First submitted 2025-01-27; First posted 2025-02-04 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-04

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhance Usual Care (Active Comparator): A sleep hygiene handout and a referral for CBT-I offered through MGH or community partners.
  Interventions: Behavioral: Enhanced Usual Care
- Survivorship Sleep Program (Experimental): 4, weekly virtual sessions of the Survivorship Sleep Program plus 1 booster session
  Interventions: Behavioral: Cognitive Behavioral Therapy - Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy - Insomnia — The Survivorship Sleep Program is a virtual program based on cognitive behavioral therapy for insomnia (CBT-I), which teaches evidence based skills to improve sleep-related behaviors, expectations, and environment, to promote relaxation, and to reduce worry. It also involves reducing the time spent in bed in order to improve the quantity and quality of sleep over time. The Survivorship Sleep Program is delivered in 4 weekly sessions by a trained facilitator and includes considerations specific to managing insomnia after cancer diagnosis and treatment. Additionally, 1 booster session is offered at week 6.
  Arms: Survivorship Sleep Program
Behavioral: Enhanced Usual Care — A sleep hygiene handout and a referral for CBT-I offered through MGH or community partners.
  Arms: Enhance Usual Care

SUMMARY:
This project is a single center, prospective randomized controlled trial (N=198) primarily evaluating the efficacy of the Survivorship Sleep Program vs. Enhanced Usual Care on insomnia severity among cancer survivors. The investigators will also examine secondary outcomes associated with cancer-related insomnia including subjective and objective sleep measures (i.e., sleep diaries, actigraphy), emotional distress, fatigue, and use of sleep medications.

Notably, most CBT-I trials with cancer survivors who have completed primary treatment with curative intent (i.e., curvivors) but not those in treatment or living with metastatic cancer (i.e., metavivors). To enhance generalizability, this RCT will stratify enrollment by survivorship phase (1:1:1).

This project in strengthened by partnerships with community organizations (SurvivorJourneys and Ellie Fund) and use of both quantitative (i.e., surveys, actigraphy) and qualitative methods (i.e., interviews) to inform considerations for future implementation.

Collectively, the proposed project will yield multiple deliverables to innovate cancer survivorship care, namely an efficacious, virtually delivered intervention addressing chronic insomnia, one of the most deleterious concerns among the growing population of cancer survivors in the US. Findings will inform a future effectiveness trial and the expansion of the synchronous delivery of CBT-I to survivors across different phases of cancer survivorship.

DETAILED DESCRIPTION:
Background: 30-50% of cancer survivors have untreated insomnia. Cognitive behavioral therapy for insomnia (CBT-I) is a first line, evidence-based treatment that is currently limited by few delivery options, lack of targeted content addressing cancer-related barriers to sleep, and limited testing by survivorship phase. With ACS pilot funding, the investigators previously developed a synchronous, virtual CBT-I program for cancer survivors (Survivorship Sleep Program; SSP) and conducted a pilot RCT demonstrating its feasibility, acceptability, and preliminary efficacy vs. enhanced usual care (EUC; CBT-I referral + sleep hygiene handout). The SSP, delivered in 6 weeks via 4 sessions + 1 booster session, is now ready for efficacy testing with a large, diverse sample including survivors who have completed primary treatment with curative intent (i.e., curvivors), survivors currently in treatment, and survivors living with metastatic cancer (i.e., metavivors).

Objective/Hypothesis: Our primary hypothesis is that the SSP (vs. EUC) will lead to significant reductions in cancer survivors' insomnia severity and secondary sleep-related outcomes.

Specific Aims: Aim 1 is to evaluate the efficacy of the SSP (vs. EUC) on the primary outcome change in insomnia severity (Insomnia Severity Index) from T0 (baseline) to T2 (4-week follow-up/10 weeks). Aim 2 is to examine changes from T0 though T3 (12-week follow-up/18 weeks) in outcomes commonly associated with cancer-related insomnia, including sleep diary and actigraphy sleep metrics (e.g., sleep efficiency), emotional distress (i.e., PROMIS depression and anxiety), daytime fatigue, use of sleep medications. Aim 3 is to characterize potential differences by cancer survivorship phase.

Study Design: The investigators propose to conduct a fully powered efficacy RCT (N=198, 1:1) evaluating the SSP (n=99) vs. EUC (n=99) among cancer survivors with insomnia. All study delivery and data collection will be conducted virtually and in close partnership with SurvivorJourneys and Ellie Fund, our community partners on this proposal. Enrollment will be stratified by 3 phases of cancer survivorship (n=66/phase, balanced between study arms). Assessments will occur at T0, T1 (6 weeks), T2, and T3. Group-by-time effects will be explicated by survivorship phase. Exit interviews assessing acceptability (enjoyableness, convenience, helpfulness, overall satisfaction) will be coded deductively (e.g., most/least) and inductively (e.g., preferences, challenges, and future delivery considerations) to extract themes by survivorship phase.

Relevance: Collectively, the proposed project will yield multiple deliverables to innovate cancer survivorship care, chiefly an efficacious, scalable, virtually-delivered intervention that addresses chronic insomnia, one of the most deleterious concerns among the growing demographic of cancer survivors in the U.S. Findings will inform a future effectiveness trial and the expansion of the synchronous delivery of CBT-I to survivors across different phases of cancer survivorship.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer survivor, defined as:

   1. (A) history of nonmetastatic, localized or regional, solid or blood malignancy(ies) and completion of primary cancer treatment (i.e., radiation, surgery, and/or chemotherapy). Use of hormonal, maintenance, oral, and immunotherapies is permitted; or
   2. (B) history of nonmetastatic, localized or regional, solid or blood malignancy(ies) and current primary cancer treatment (i.e., radiation, surgery, and/or chemotherapy); Use of hormonal, maintenance, oral, and immunotherapies is permitted; or
   3. (C) history of metastatic sold or blood malignancy (ies) taking hormonal, maintenance, oral, or immunotherapies to prevent further disease progression.
2. Chronic insomnia (DSM-5 criteria)
3. Age 18 years or older

Exclusion Criteria:

1. Self-reported inability to speak and write in English
2. Undertreated non-insomnia sleep disorder (e.g., sleep apnea)
3. Undertreated epilepsy, undertreated serious mental illness, undertreated suicidality, and/or psychiatric hospitalization in the past year
4. Unwilling or unable to discontinue night shift work

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | Screening, baseline, week 6, week 10, and week 18
  A 7-item self-report questionnaire measuring changes in insomnia severity. Response options range from 0 (None) to 4 (Very severe). Items include "How NOTICEABLE to others do you think your sleep problem is in terms of impairing the quality of your life?"

SECONDARY OUTCOMES:
PROMIS anxiety short form | Baseline, Week 6, week 10, and week 18
  A 4-iem self-report questionnaire measuring anxiety levels. Response options range from 1 (Never characteristic of me in the past seven days) to 5 (Always as it applies within the past seven days). Items include "In the past seven days I felt fearful" and "In the past seven days I felt anxious."
PROMIS depression short form | Baseline, week 6, week 10, and week 18
  A 4-iem self-report questionnaire measuring depression levels. Response options range from 1 (Never characteristic of me in the past seven days) to 5 (Always as it applies within the past seven days). Items include "In the past seven days I felt worthless" and "In the past seven days I felt unhappy."
PROMIS fatigue short form | baseline, week 6, week 10, and week 18
  A 7-iem self-report questionnaire measuring fatigue levels. Response options range from 1 (Never characteristic of me in the past seven days) to 5 (Always as it applies within the past seven days). Items include "In the past seven days, how often did you feel tired?" and "In the past seven days, how often did you run out of energy?"
Use of sleep aid meditations | baseline, week 6, week 10, and week 18
  Use of sleep aid medications (frequency, dose) will be evaluated via self-report surveys and electronic medical records (when possible).
Perceived Cognitive Impairment subscale of The Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) | baseline, week 6, week 10, and week 18
  A 20-item questionnaire measuring perceived cognitive impairments. Responses range from 0, ''never,'' to 4, ''several times a day,'' in the previous 7 days and negatively worded items are reverse scored to create subscale scores. Items include "My thinking has been slow."
Sleep diaries and actigraphy/Fitbit | baseline, week 6, week 10, and week 18
  Sleep diaries and actigraphy/Fitbit will be collected during SSP Sessions 1-4 and for 7 days at each timepoint (T0-T3) to derive sleep efficiency, sleep onset latency, and wake after sleep onset. Discrepancy scores between subjective and objective sleep metrics (e.g., sleep onset latency) will be examined. Participants will be asked to wear sleep tracking devices (actigraphs/Fitbit) to objectively assess their sleep. These devices will be mailed to participants along with detailed instructions about when and how to wear the devices. Study participants will mail back the devices to the study team upon completion of data collection. All devices will be thoroughly disinfected by study staff between usages to prevent the spread of disease. Importantly, wearing an actigraph/Fitbit is optional, participants may participate in the study if they do not wish to be included in this study component.
Smoking | baseline, week 6, week 10, and week 18
  A 2-item self-report questionnaire measuring current and prior cigarette smoking status. Items include, "Do you now smoke cigarettes every day, some days, or not at all?" and "About how long has it been since you last smoked a cigarette, even a puff?
International Physical Activity Questionnaire | baseline, week 6, week 10, and week 18
  A 4-item self-report questionnaire measuring physical activity in the past 7 days. Items include, "on how many days did you do vigorous physical activities like heavy lifting, digging, aerobics, or fast bicycling?".
Perceived weight changes | baseline, week 6, week 10, and week 18
  A 2-item self-report questionnaire assessing accidental weight changes as a result of cancer treatment and intentional weight changes.
Fear of Cancer Recurrence Inventory-Severity subscale | baseline, week 6, week 10, and week 18
  FCR severity is assessed using the FCR Inventory severity subscale (range 0-36, 16=elevated FCR; 22=clinically elevated FCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States